CLINICAL TRIAL: NCT00736398
Title: Fusion Assessment Clinical Trial (FACT)
Brief Title: Fusion Assessment Clinical Trial
Acronym: FACT
Status: Completed | Type: Observational
Sponsor: Flexuspine, Inc. (Industry)
Responsible Party: Vin Jannetty / CEO, Flexuspine, Inc.
Other Study IDs: 01000-T02
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Spinal Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Spinal fusion
  Interventions: Procedure: Spinal fusion

INTERVENTIONS:
Procedure: Spinal fusion — Spinal fusion

SUMMARY:
This is an observational study to assess clinical outcomes in patients who undergo spinal fusion. Patients who are already scheduled for spinal fusion will enroll in the study. Information about prior therapies will be collected, and then patients will be followed to see how they do after spinal fusion. This study will help researchers better understand the natural course of patients who patients who undergo spinal fusion surgery.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar DDD
* Candidate for spinal fusion
* Provide written informed consent

Exclusion Criteria:

* Prior lumbar spinal fusion
* Metabolic bone disease
* Morbid obesity
* Systemic infection or active malignancy
* Pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring spinal fusion
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-08

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Florida Spine Institute, Clearwater, Florida
  - Foundation for Orthopaedic Research and Education, Temple Terrace, Florida
  - Greater Baltimore Medica Center, Baltimore, Maryland
  - The Washington Hospital, Washington, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Guy Danielson, M.D., Tyler, Texas